CLINICAL TRIAL: NCT06880094
Title: Study of Congenital Orofacial Clefts by Implementing Optical Genome Mapping
Acronym: CARTOFENTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2023_843_0023
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Orofacial Clefts; Next Generation Sequencing (NGS); Optical Genome Mapping
Keywords: orofacial clefts; Next Generation Sequencing; Optical Genome Mapping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with syndromic, familial or complex orofacial clefts (Experimental)
  Interventions: Genetic: blood withdrawal

INTERVENTIONS:
Genetic: blood withdrawal — blood withdrawal for genetic testing

SUMMARY:
Orofacial clefts, the most common congenital craniofacial malformations, have a complex etiology involving an interaction between genetic and environmental factors.

Chromosomal abnormalities, including structural variations, represent a major cause of human pathology. Recently, technological developments and the introduction of next-generation sequencing (NGS) technologies have revolutionized the field of medical genetics.

Optical genome mapping (OGM) is an innovative, high-resolution "long read" technique that enables the identification of all classes of chromosomal variation, consisting in the direct visualization of long, labeled DNA molecules throughout the genome. This technology is gradually becoming an essential tool for studying onco-hematology and constitutional genetic pathologies The purpose of this study is to search for structural chromosomal variants (SV) or copy number variants (CNV) not identifiable either by cytogenetic methods nor by "short read" NGS "short read, in individuals with oral-facial clefts with no genetic diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with syndromic, complex or familial oral-facial clefts
* With no established genetic diagnosis
* Followed up at the Amiens-Picardie University Hospital

Exclusion Criteria:

* genetic diagnosis of oral-facial cleft
* No health insurance affiliation
* Patient under guardianship or curatorship, under safeguard of justice or deprived under public law
* Pregnant, parturient or breast-feeding woman

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Identification of a structural chromosomal variant | 2 years
  Identification of a structural chromosomal variant involved in the genesis of orofacial clefts by studying the genetic characteristics of individuals with orofacial clefts.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No